CLINICAL TRIAL: NCT03747757
Title: Cognitive Behavioral Therapy (CBT) Intervention for Cancer Related Fatigue (CRF) in Patients With AML and Lymphoma
Brief Title: Cognitive Behavioral Therapy in Helping Patients With Acute Myeloid Leukemia or Lymphoma With Cancer-Related Fatigue
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0542; NCI-2018-02528 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0542 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2018-11-15; First posted 2018-11-20 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Cancer Fatigue; Lymphoma; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Lymphoma | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (CBT) (Experimental): Patients undergo CBT consisting of 7 counseling sessions, up to 45 minutes each over the phone.
  Interventions: Behavioral: Cognitive Behavior Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy — Undergo CBT
  Other Names: CBT; cognitive therapy; CT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well cognitive behavioral therapy works in helping patients with acute myeloid leukemia or lymphoma with cancer-related fatigue. Behavioral therapy uses methods to help patients change the way they think and act. Behavioral skills may help patients with acute myeloid leukemia or lymphoma cope with anxiety, depression, and other factors that may influence their level of cancer-related fatigue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether acute myeloid leukemia (AML) and lymphoma patients with cancer-related fatigue (CRF) will be satisfied with the cognitive behavioral therapy (CBT) intervention, and if CBT will be feasible for AML and lymphoma patients with CRF where the feasibility will be based on adherence measurement.

SECONDARY OBJECTIVES:

I. To examine the preliminary effects of CBT on improvement of CRF (Functional Assessment of Cancer Illness Therapy (FACIT-F) - Fatigue subscale, its related symptoms, M.D. Anderson Symptom Inventory - Acute Myeloid Leukemia / Myelodysplastic Syndromes (MDASI-AML/MDS), Pittsburgh Sleep Quality Index (PSQI), Hospital Anxiety Depression Scale (HADS), and Quality of Life (FACT-G) in AML and lymphoma patients receiving this combination regimen at the end of 8 weeks or 6 months.

EXPLORATORY OBJECTIVES:

I. To explore the effects of CBT on hope for future and burdens of treatment and their interference with patients' lives using the Herth Hope Index (HHI), and MDASI-AML/MDS.

OUTLINE:

Patients undergo CBT consisting of 7 counseling sessions, up to 45 minutes each over the phone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML or AML secondary to MDS (myelodysplastic syndrome) and lymphoma with fatigue >= 4/10 (0-10 scale) on the MDASI-AML/MDS.
* Presence of fatigue for at least 2 weeks.
* Normal cognition by Memorial Delirium Assessment Scale score of < 13 at baseline.
* Hemoglobin > 8 g/L within 2 weeks of enrollment in the study; if the patient has not had blood drawn for a hemoglobin level in the past two weeks, one will be done to determine the eligibility.
* Zubrod performance status =< 2.
* Able to communicate in English or Spanish.
* Seen at leukemia and lymphoma clinics at University of Texas (UT) MD Anderson Cancer Center, Houston, Texas and its affiliates in University of Texas.

Exclusion Criteria:

* Has received CBT (cognitive behavioral therapy) for any indication (e.g. depression, sleep disturbance) in the past 1 year.
* Inability to comply with study protocol procedures.
* Prior cancer diagnosis other than noted in the inclusion criterion #1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2027-09-11 (Estimated); Study Completion 2027-09-11 (Estimated)

PRIMARY OUTCOMES:
Adherence to cognitive behavioral therapy (CBT) defined as percentage of the total completed prescribed counseling sessions (7 sessions) the study patient is able to complete | Up to 8 weeks or 6 months
Satisfaction with CBT assessed using a 5 point, fully word-anchored balanced bipolar scale (Satisfaction Assessment). | Up to 8 weeks
  To determine if patients are satisfied with CBT, based on equal to or more than 75% of patients indicating their satisfaction with CBT with a rating of "somewhat satisfied" or "completely satisfied". Satisfaction will be assessed using a 5 point, fully word-anchored balanced bipolar scale (Satisfaction Assessment).

SECONDARY OUTCOMES:
Improvement of symptoms determined by M.D. Anderson Symptom Inventory - Acute Myeloid Leukemia / Myelodysplastic Syndromes (MDASI-AML/MDS) | Baseline to 8 weeks or 6 months
  MDASI symptom questionnaire answers range from 0 meaning "Not Present" to 10 meaning "As Bad as You Can Imagine".

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Yennu, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Yennurajalingam S, Konopleva M, Carmack CL, Dinardo CD, Gaffney M, Michener HK, Lu Z, Stanton P, Ning J, Qiao W, Bruera E. Treatment of Cancer-related-Fatigue in Acute Hematological Malignancies: Results of a Feasibility Study of using Cognitive Behavioral Therapy. J Pain Symptom Manage. 2023 Mar;65(3):e189-e197. doi: 10.1016/j.jpainsymman.2022.11.003. Epub 2022 Nov 13. PMID 36384181
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org